CLINICAL TRIAL: NCT02300415
Title: Comparison of Sensitivity Between Presepsine and Arterial Lactate for the Diagnosis of Severe Sepsis and Sepsis Shock in Emergency Department.
Brief Title: Comparison of Sensitivity Between Presepsine and Lactate for the Diagnosis of Severe Sepsis.
Acronym: PREDI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 14-PP-15
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Severe Sepsis and Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — total blood sample

GROUPS / COHORTS (1):
- patient with sepsis: Patients admitted to the emergency department and with criteria of sepsis.
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — Dosage of presepsine

SUMMARY:
Severe sepsis and sepsis shock are common in emergency department, with a high mortality rate. The potential severity of this disease impose a diagnosis as early as possible to start antibiotic therapy and hemodynamic support. Conventional biomarkers are an important support for the emergency physician. However, comparison of sensitivity and specificity for new biomarkers, like presepsine, suggests that they can be more efficient in this area.

In this single-center, prospective, non-interventional study, we propose to compare the sensitivity of presepsine to that of lactate for the diagnosis of severe sepsis and septic shock We emit to main hypothesis that the sensitivity of presepsine is higher than that of lactate for the diagnosis of severe sepsis.

DETAILED DESCRIPTION:
Severe sepsis and sepsis shock are common in emergency department, with a high mortality rate. The potential severity of this disease impose a diagnosis as early as possible to start antibiotic therapy and hemodynamic support. The conventional biomarkers are an important support for the emergency physician. However, comparison of sensitivity and specificity for new biomarkers, like presepsine, suggest that they can be more efficient in this indication. Presepsine is a soluble fragment of CD14, its concentration is a reflection of cellular activity (macrophages and monocytes) in response of a sepsis's aggression. Today, it's possible to asses the presepsine value at bedside, with new device (PATHFAST), in just 17 minutes, reinforcing the interest for this biomarker.

We will conduct a single-center, prospective, non-interventional study, between december 2014 and July 2015 in the university emergency department of Nice. The primary outcome is to compare the sensitivity of presepsine to lactate for the diagnosis of severe sepsis and septic shock. The dosage of presepsine will be made in 194 patients over 18 years old , with at least two S.I.R.S criteria, a suspected infection, and the presence of one organ failure.

The secondary outcomes are to asses the link between the presepsine value and the germ responsible of sepsis, the correlation between presepsine value at the admission and the mortality at J-28. And we will try to determine if there is a correlation between the initial presepsine value, and the P.I.R.O score.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Presence of at least two SIRS criteria (T °> 38.3 ° or <36 °, tachycardia> 90 / min, tachypnea> 20 / min, recent alteration of consciousness)
* Suspected Infection
* Indication of an arterial lactate assay on medical advice
* Affiliation to social security
* Informed Consent

Exclusion Criteria:

* Renal dialysis
* Scalable neoplasia chemotherapy
* Patient Palliative Care
* Private Patient freedom or under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with septic shock or severe sepsis
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Presepsine and lactate values | Day 0
  Presepsine and lactate values at the admission in ED for the patients with severe sepsis criteria

SECONDARY OUTCOMES:
Sepsis shock | Day 0
  Sepsis shock. (Sepsis shock will be defined if blood pressure is < 90mmhg after fluid resuscitation or if catecholamine is used)
Mortality | Day 28
  Mortality at J-28
Germs responsible of sepsis | Day 0
  Type of germs responsible of sepsis (found on blood culture in emergency department)
PIRO Score | Day 0
  P.I.R.O score at the admission in ED

CONTACTS AND LOCATIONS:
Overall Officials: Julie CONTENTI, PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France